CLINICAL TRIAL: NCT06513052
Title: Effect of Consuming Flavanol-rich Cocoa on Biomarkers Associated with Digestive and Cerebrovascular Health in the Colombian Adult Population
Brief Title: Flavanol-rich Cocoa on Digestive and Cerebrovascular Health in the Colombian Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vidarium, Nutrition, Health and Wellness Research Center (Other)
Collaborators: CES University (Other); Compañia Nacional de Chocolates (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CF-2024
Record Dates: First submitted 2024-07-12; First posted 2024-07-22 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Cocoa flavanols; Gut-brain axis; Gut microbiota; Vascular function; Gastrointestinal health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): <100 mg cocoa flavanols/day for 12 weeks
  Interventions: Other: Commercial cocoa
- Intervention (Experimental): 500 mg cocoa flavanols/day for 12 weeks
  Interventions: Other: High flavonols Cocoa

INTERVENTIONS:
Other: Commercial cocoa — daily intake of a beverage made with 8 grams of commercial cocoa low in flavanols, dissolved in 200 mL of low-fat, lactose-free milk
  Arms: Control
Other: High flavonols Cocoa — Daily intake of a beverage made with 8 grams of cocoa high in flavanols, dissolved in 200 mL of low-fat, lactose-free milk.
  Arms: Intervention

SUMMARY:
The purpose of this study is to investigate the effects of consuming flavanol-rich cocoa on biomarkers associated with digestive and cerebrovascular health in a group of adults.

DETAILED DESCRIPTION:
The study seeks 40 adults aged 20-50 with normal or slightly overweight (by BMI) who regularly consume cocoa/chocolate. After recruitment, participants will receive a detailed explanation of the objectives and conditions of the study and will sign the informed consent and will be randomly assigned to randomly divided into two groups: Control Group that consumes a daily beverage with low-flavanol cocoa or the intervention group that consumes a daily beverage with high-flavanol cocoa. Participants in each intervention arm will be matched by BMI category (normal weight or overweight), sex (female or male), and age (plus or minus 5 years). Both groups will consume a single daily serving (8 grams) of their assigned cocoa (packaged individually) dissolved in low-fat and lactose-free milk (200 ml) before or with their breakfast. At baseline (time 0) and at the end of the intervention (12 weeks), each participant will be assessed for biological indicators gastrointestinal health, the composition of the gut microbiota and cerebrovascular health, markers associated with neuroinflammation, oxidative stress, and barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 50 years.
* Participants should be regular consumers of either table chocolate or cocoa powder
* Participants should have a BMI within the normal range, which is typically between 18.5 and 24.9 kg/m2. Overweight individuals with a BMI between 25 and 27 kg/m2 may also be eligible. (have a BMI within the normal or slightly overweight range)

Exclusion Criteria:

* Individuals who experience intolerance or adverse effects to the study products during the intervention period will be withdrawn from the trial
* Participants who become pregnant during the study will be excluded.
* Individuals who are diagnosed with Gastrointestinal diseases: This includes liver disorders, duodenal ulcers, gastritis, malabsorption disorders, short bowel syndrome, diverticulosis, Crohn's disease, ulcerative colitis, irritable bowel syndrome, and celiac disease. Central nervous system diseases: This includes vascular dementia and other neurodegenerative diseases. Inflammatory diseases, Malignant neoplasms, Diabetes mellitus, Cardiovascular diseases and Recent fractures.
* Significant alcohol consumption: Participants who consume more than 1 alcoholic drink per day for women or 2 alcoholic drinks per day for men.
* High coffee consumption: Participants who consume more than 2 cups of coffee per day will be excluded.
* Regular use of certain medications: Participants who regularly consume (within the past 3 months) any of the following medications: Metformin, Steroid anti-inflammatory drugs (NSAIDs) like dexamethasone, prednisone, triamcinolone, prednisolone, betamethasone, hydrocortisone, deflazacort, paramethasone, and fludrocortisone. Proton pump inhibitors (PPIs) like omeprazole, esomeprazole, lansoprazole, rabeprazole, pantoprazole, and dexlansoprazole. Hypnotic medications: These include drugs like zolpidem, zaleplon, alprazolam, diazepam, lorazepam, midazolam, and flurazepam. Antibiotics, antiparasitics, or laxatives. Medications containing acetylsalicylic acid (aspirin) or 5-alpha reductase inhibitors (finasteride, dutasteride).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-01-26 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal health | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in Gastrointestinal Symptom Assessment Scale (GSRS) scores. The GSRS is a 7-point scale ranging from 1 (no discomfort at all) to 7 (severe discomfort), with higher scores indicating worse gastrointestinal symptoms.
Gut microbiota composition | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in the Abundance of the beneficial bacteria Bifidobacterium and Lactobacillus, as well as opportunistic pathogens belonging to the Enterobacteriaceae family.
Vascular function | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of Endothelin-1 in pg/ml

SECONDARY OUTCOMES:
Blood pressure | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in systolic and diastolic blood pressure in mm Hg
Blood lipid profile | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in serum levels of total cholesterol in mg/dL, LDL cholesterol in mg/dL, HDL cholesterol in mg/dL and triglycerides in mg/dL.
Glucose metabolism | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in fasting blood glucose levels in mg/dL
Markers associated with neuroinflammation | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of interleukin 6 (IL-6) in pg/mL, and tumor necrosis factor alpha (TNF-α) in pg/mL
Markers associated with systemic inflammation | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of high sensitivity C reactive protein (hsCRP) in mg/L
Markers associated with oxidative stress | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in urine levels of 8-isoprostane corrected for creatinine clearance (ng/mg creatinine).
  Corrected urine 8-isoprostane levels will be calculated by dividing urine 8-isoprostane levels in ng/ml by urine creatinine levels in mg/ml.
Other markers associated with oxidative stress | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma oxysterol levels in µg/ml
Markers associated with Barrier function | At baseline (time 0) and at the end of the intervention (12 weeks)
  Plasma levels of Lipopolysaccharide-binding protein (LBP) in ng/ml, neuron-specific enolase (NSE) in ng/ml and neuregulin-1β in ng/ml.
Markers associated with angiogenesis | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of Vascular Endothelial Growth Factor (VEGF) in pg/ml
Markers associated with endothelial function | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of endocan in ng/ml, and endostatin in ng/ml
Other markers associated with endothelial function | At baseline (time 0) and at the end of the intervention (12 weeks)
  Changes in plasma levels of nitric oxide (NO) in micromol per liter (µM)

CONTACTS AND LOCATIONS:
Overall Officials: Jelver Sierra, PhD, Principal Investigator — Vidarium, Nutrition, Health and Wellness Research Center
Locations (1):
- Vidarium, Nutrition, Health and Wellness Research Center, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
The data will be available when the results are published. The data can be obtained by downloading from the cloud (ex: Sequence Read Archive data at National center for biotechnology information (NCBI-SRA) or GitHub)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available when the results are published.
Access Criteria: Public